CLINICAL TRIAL: NCT01986530
Title: Circulating Irisin in Healthy Young Men and Women and Correlation With Lean Body Mass, Fat Mass and Adipocytokines. Circadian and Seasonal Variation and the Effect of Food Intake and Exercise
Brief Title: Circulating Levels of Irisin in Healthy Young Subjects
Acronym: IRISSAS
Status: Completed | Type: Observational
Sponsor: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Athanasios D. Anastasilakis, Consultant of Endocrinology, 424 General Military Hospital
Other Study IDs: SSAS-1-MANTZ; 424-IRIS (Other: 424MHTH-1453/28-01-13)
Record Dates: First submitted 2013-11-09; First posted 2013-11-18 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Subjects
Keywords: irisin; adiponectin; leptin; lean body mass; fat mass
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Healthy individuals: Participants will be healthy volunteers of both sexes recruited from the Greek Military Medical School personnel, Thessaloniki, Greece.
- Boost Subgroup: After an overnight fast, 40 participants will be provided a standardized mixed meal in two different quantities (125 ml, n=20 and 250 ml, n=20) and blood samples will be obtained before as well as 30 min after mixed meal ingestion
  Interventions: Dietary Supplement: Boost
- Aerobic exercise: After an overnight fast, 20 participants will be subjected to aerobic exercise for 30 min and blood samples will be obtained at baseline and at 30 min
  Interventions: Other: Aerobic exercise
- Circadian variation Subgroup: 20 of the participants will be hospitalized and closely monitored for 24 hours. A catheter will be inserted in a vein and blood samples will be obtained every 3 hours through the 24-hour period.
- Seasonal variation Subgroup: 20 of the participants will be monitored for one year and blood samples will be obtained every 3 months (at the middle of month January - April - July - October). Subjects will be instructed to maintain their normal exercise routine and dietary habits.

INTERVENTIONS:
Dietary Supplement: Boost — After an overnight fast, blood samples will be obtained before as well as 30 min after standardized mixed meal ingestion
  Groups: Boost Subgroup
Other: Aerobic exercise — After an overnight fast and rest, blood samples will be obtained before as well as 30 min after aerobic exercise
  Groups: Aerobic exercise

SUMMARY:
Irisin, a newly discovered myokine induced in exercise, has potential effects in stimulating adipose tissue browning, fighting obesity and diabetes. No prior study has reported on the role of circulating irisin in healthy individuals in correlation with lean and fat body mass. Furthermore, the circadian and seasonal variation of irisin is largely unknown.

DETAILED DESCRIPTION:
The main aims of this prospective study will be to investigate: 1) circulating irisin levels in healthy, young men and women according to their lean and fat mass; 2) the circadian variations of irisin levels; 3) the seasonal variations of irisin levels.

ELIGIBILITY:
Inclusion Criteria: Healthy volunteers

Exclusion Criteria: i) body mass index (BMI) above 30 or below 20 kg/m2; ii) diseases that could affect muscle or fat homeostasis; iii) medications that could affect muscle or fat homeostasis.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be healthy volunteers of both sexes recruited from the Greek Military Medical School personnel, Thessaloniki, Greece.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Irisin | 1 day
  After a standardized dinner and an overnight fast, a blood sample will be obtained the next morning.
irisin circadian variation | 1 day
  20 participants will be hospitalized and closely monitored for 24 hours. A catheter will be inserted in a vein and blood samples will be obtained every 3 hours through the 24-hour period
irisin seasonal variation | 12 months
  20 participants will be monitored for one year and blood samples will be obtained every 3 months (at the middle of month January - April - July - October). At the same intervals physical examination and BMI calculation will be conducted. Subjects will be instructed to maintain their normal exercise routine and dietary habits.
Irisin postprandial | 1 day
  A sub-population of 40 participants of the cohort will receive a standardized meal (Boost) in two different quantities (20 participants will receive 125 ml and 20 participants 250 ml). Serum irisin levels will be measured at baseline and 30 min postprandial.
Irisin after excercise | 1 day
  A sub-population of 20 participants of the cohort will be subjected to 30 min of aerobic exercise. Serum irisin levels will be measured at baseline and at 30 min.

SECONDARY OUTCOMES:
Irisin associates | 1 day
  After a standardized dinner and an overnight fast, a blood sample for adiponectin and leptin will be obtained the next morning, and body composition (total body fat mass and bone-free lean mass) will be assessed by BIA. Participants will also be asked to complete a validated questionnaire assessing their diet and exercise habits. Correlations between serum irisin levels and the above parameters will be examined
serum adipokines | 1 day
  After a standardized dinner and an overnight fast, a blood sample for adiponectin and leptin will be obtained the next morning.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios D Anastasilakis, MD, PhD, Principal Investigator — 424 General Military Hospital
Locations (1):
- 424 General Military Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Polyzos SA, Kountouras J, Anastasilakis AD, Geladari EV, Mantzoros CS. Irisin in patients with nonalcoholic fatty liver disease. Metabolism. 2014 Feb;63(2):207-17. doi: 10.1016/j.metabol.2013.09.013. Epub 2013 Oct 18. PMID 24140091
- [Background] Vamvini MT, Aronis KN, Panagiotou G, Huh JY, Chamberland JP, Brinkoetter MT, Petrou M, Christophi CA, Kales SN, Christiani DC, Mantzoros CS. Irisin mRNA and circulating levels in relation to other myokines in healthy and morbidly obese humans. Eur J Endocrinol. 2013 Oct 21;169(6):829-34. doi: 10.1530/EJE-13-0276. Print 2013 Dec. PMID 24062354
- [Background] Polyzos SA, Kountouras J, Shields K, Mantzoros CS. Irisin: a renaissance in metabolism? Metabolism. 2013 Aug;62(8):1037-44. doi: 10.1016/j.metabol.2013.04.008. Epub 2013 May 10. No abstract available. PMID 23664085
- [Background] Huh JY, Panagiotou G, Mougios V, Brinkoetter M, Vamvini MT, Schneider BE, Mantzoros CS. FNDC5 and irisin in humans: I. Predictors of circulating concentrations in serum and plasma and II. mRNA expression and circulating concentrations in response to weight loss and exercise. Metabolism. 2012 Dec;61(12):1725-38. doi: 10.1016/j.metabol.2012.09.002. Epub 2012 Sep 25. PMID 23018146
- [Derived] Anastasilakis AD, Polyzos SA, Saridakis ZG, Kynigopoulos G, Skouvaklidou EC, Molyvas D, Vasiloglou MF, Apostolou A, Karagiozoglou-Lampoudi T, Siopi A, Mougios V, Chatzistavridis P, Panagiotou G, Filippaios A, Delaroudis S, Mantzoros CS. Circulating irisin in healthy, young individuals: day-night rhythm, effects of food intake and exercise, and associations with gender, physical activity, diet, and body composition. J Clin Endocrinol Metab. 2014 Sep;99(9):3247-55. doi: 10.1210/jc.2014-1367. Epub 2014 Jun 10. PMID 24915120